CLINICAL TRIAL: NCT01708915
Title: A Multi-centre, Double-blind, Randomised, Parallel Group Study to Assess the Efficacy and Safety of Multiple Doses of Topically Applied Hyperemisation-inducing Ointment (2cm Ointment Line Per Application; up to 3 Times Daily for up to 4 Days) Containing 2.5% Nicoboxil/0.4% Nonivamide Versus 2.5% Nicoboxil, 0.4% Nonivamide and Placebo in Patients 18 to 65 Years of Age With Acute Low Back Pain
Brief Title: Nonivamide/Nicoboxil Ointment in Acute Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 69.52; 2011-003890-27 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-10-16; First posted 2012-10-17 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2014-05-29 (Estimated); Status verified 2014-05

CONDITIONS: Acute Low Back Pain
MeSH Terms: interventions — nicoboxil; nonivamide

ARMS (4):
- nonivamide + nicoboxil (Finalgon) (Active Comparator): 2cm ointment line for a skin area of approximately 20 cm x 20 cm up to 3 times in a 24h period
  Interventions: Drug: nonivamide + nicoboxil (Finalgon)
- nonivamide (Active Comparator): 2cm ointment line for a skin area of approximately 20 cm x 20 cm up to 3 times in a 24h period
  Interventions: Drug: nonivamide
- nicoboxil (Active Comparator): 2cm ointment line for a skin area of approximately 20 cm x 20 cm up to 3 times in a 24h period
  Interventions: Drug: nicoboxil
- placebo (Placebo Comparator): 2cm ointment line for a skin area of approximately 20 cm x 20 cm up to 3 times in a 24h period
  Interventions: Drug: placebo matching nonivamide + nicoboxil

INTERVENTIONS:
Drug: nicoboxil — 2cm ointment line for a skin area of approximately 20 cm x 20 cm up to 3 times in a 24h period
  Arms: nicoboxil
Drug: placebo matching nonivamide + nicoboxil — 2cm ointment line for a skin area of approximately 20 cm x 20 cm up to 3 times in a 24h period
  Arms: placebo
Drug: nonivamide + nicoboxil (Finalgon) — 2cm ointment line for a skin area of approximately 20 cm x 20 cm up to 3 times in a 24h period
  Arms: nonivamide + nicoboxil (Finalgon)
Drug: nonivamide — 2cm ointment line for a skin area of approximately 20 cm x 20 cm up to 3 times in a 24h period
  Arms: nonivamide

SUMMARY:
The aim of this study is to assess the efficacy and tolerability of Nicoboxil/Nonivamide ointment in comparison to Nicoboxil, Nonivamide, and placebo ointments for the treatment of acute low back pain.

ELIGIBILITY:
Inclusion criteria:

* Patients must sign and date an Informed Consent consistent with International Conference on Hermonisation (ICH)/Good Clinical Practice (GCP) guidelines and local regulation prior to participation in the trial.
* Patients must agree to cooperate with all trial evaluations and perform all required tasks.
* Acute low back pain for more than 2 days and less than 21 days (= 3 weeks)
* Male or female patients aged 18 to 65 years
* Low back pain rating >5 on a 0-10 numerical rating scale (NRS).
* Female patients of childbearing potential may participate only in case of availability of a negative urine pregnancy test and a confirmed menstrual period prior to study entry and using a highly effective method of birth control. Highly effective methods of birth control are defined as those which result in a low failure rate (i.e. less than 1 % per year) when used consistently and correctly such as implants, injectables, combined oral contraceptives, appropriate intrauterine devices, sexual abstinence or vasectomised partner. Barrier methods of contraception (e.g. condom, diaphragma or occlusive cap) are accepted if used in combination with spermicides (e.g. foam, gel). Female patients will be considered being of childbearing potential unless surgically sterilised by bilateral tubal ligation/salpingectomy or hysterectomy or post-menopausal for at least one year.

Exclusion criteria:

* Multilocular pain or panalgesia
* History of more than three low back pain episodes in the last six months
* Abnormal findings in at least one of the following assessments: Achilles tendon reflex, patella reflex, heel walking, toe walking, cutaneous sensitivity of the legs (including gluteal region), paresis tests in supine position upon dorsiflexion, plantarflexion, hip flexion, knee extension
* Bladder and/or rectum dysfunction
* Acute low back pain due to vertebral collapse or neoplastic, inflammatory (ankylosing spondylitis), traumatic, or infective origins
* Any condition, disease or concomitant treatment that in the judgement of the Investigator will affect the subject's ability to participate in the clinical trial or which will influence the test methodology used
* Negative experience in the past with heat treatment for muscle complaints (e. g. hot water bottle, heat pads, hyperemisation-inducing topical creams, ointments or patches)
* History of treatment of back pain with centrally acting analgesics (e. g. opioids) and muscle relaxants
* Surgery due to back pain or rehabilitation due to back pain in the last 12 months
* Spinal injection back pain treatment within 6 months prior to enrollment
* Intake of antidepressant/antipsychotic medication within 4 weeks prior to enrollment
* Treatment of the recent low back pain period with oral analgesics for more than 4 consecutive days
* Locally applied medication to the back within 48 hours prior to enrollment (topical treatments, injections)
* Administration of other analgesics within 24 h prior to enrollment (exception: acetyl salicylic acid (ASS) up to 100 mg/daily for anti platelet-aggregation therapy)
* Non-pharmacological low back pain treatment (physiotherapy, heat treatment (e.g. hot water bottle, heat patch, or massages) within 12 h prior to enrollment
* Participation in an investigational drug or device trial within 4 weeks prior to enrollment
* Hypersensitivity to Nicoboxil, Nonivamide, or paracetamol
* Known hypersensitivity to any other ingredient, especially to sorbic acid/sorbate, to citronella oil containing e.g. the fragrance compounds geraniol, citronellol and citronellal, or to relevant flowers containing these compounds such as geranium, lavender, jasmine or rose. For patients with known hypersensitivity to perfumes or known type IV hypersensitivity to fragrance-mix I, the application of the investigational product should be performed only with particular caution.
* Skin lesions (e. g., rash, dermatitis, bruising, laceration) in the back region
* Drug dependence and/or alcohol abuse
* Severe hepatocellular insufficiency
* Patients who are pregnant or breast-feeding

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 805 (Actual)
Dates: Start 2012-10; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (37):
- Germany (37):
  - 69.52.49007 Boehringer Ingelheim Investigational Site, Bad Lippspringe
  - 69.52.49003 Boehringer Ingelheim Investigational Site, Berlin
  - 69.52.49004 Boehringer Ingelheim Investigational Site, Berlin
  - 69.52.49026 Boehringer Ingelheim Investigational Site, Berlin
  - 69.52.49032 Boehringer Ingelheim Investigational Site, Berlin
  - 69.52.49033 Boehringer Ingelheim Investigational Site, Berlin
  - 69.52.49041 Boehringer Ingelheim Investigational Site, Berlin
  - 69.52.49027 Boehringer Ingelheim Investigational Site, Cologne
  - 69.52.49035 Boehringer Ingelheim Investigational Site, Cologne
  - 69.52.49040 Boehringer Ingelheim Investigational Site, Cologne
  - 69.52.49002 Boehringer Ingelheim Investigational Site, Einbeck
  - 69.52.49024 Boehringer Ingelheim Investigational Site, Essen
  - 69.52.49031 Boehringer Ingelheim Investigational Site, Essen
  - 69.52.49036 Boehringer Ingelheim Investigational Site, Essen
  - 69.52.49005 Boehringer Ingelheim Investigational Site, Everswinkel
  - 69.52.49039 Boehringer Ingelheim Investigational Site, Fürth
  - 69.52.49018 Boehringer Ingelheim Investigational Site, Goch
  - 69.52.49025 Boehringer Ingelheim Investigational Site, Großheirath-Rossach
  - 69.52.49022 Boehringer Ingelheim Investigational Site, Haag
  - 69.52.49009 Boehringer Ingelheim Investigational Site, Hamburg
  - 69.52.49019 Boehringer Ingelheim Investigational Site, Hamburg
  - 69.52.49015 Boehringer Ingelheim Investigational Site, Kaarst
  - 69.52.49042 Boehringer Ingelheim Investigational Site, Karlsruhe-Rüppurr
  - 69.52.49013 Boehringer Ingelheim Investigational Site, Köthen
  - 69.52.49014 Boehringer Ingelheim Investigational Site, Künzing
  - 69.52.49034 Boehringer Ingelheim Investigational Site, Ludwigshafen
  - 69.52.49028 Boehringer Ingelheim Investigational Site, Messkirch
  - 69.52.49030 Boehringer Ingelheim Investigational Site, Messkirch
  - 69.52.49029 Boehringer Ingelheim Investigational Site, Münster
  - 69.52.49012 Boehringer Ingelheim Investigational Site, Neunkirchen
  - 69.52.49020 Boehringer Ingelheim Investigational Site, Rodgau
  - 69.52.49037 Boehringer Ingelheim Investigational Site, Siegen
  - 69.52.49016 Boehringer Ingelheim Investigational Site, Stockach
  - 69.52.49010 Boehringer Ingelheim Investigational Site, Straßkirchen
  - 69.52.49021 Boehringer Ingelheim Investigational Site, Villingen-Schwenningen
  - 69.52.49023 Boehringer Ingelheim Investigational Site, Wangen
  - 69.52.49011 Boehringer Ingelheim Investigational Site, Weilburg

REFERENCES:
- [Derived] Gaubitz M, Schiffer T, Holm C, Richter E, Pisternick-Ruf W, Weiser T. Efficacy and safety of nicoboxil/nonivamide ointment for the treatment of acute pain in the low back - A randomized, controlled trial. Eur J Pain. 2016 Feb;20(2):263-73. doi: 10.1002/ejp.719. Epub 2015 Apr 30. PMID 25929250

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Patients treated with placebo ointment
- Nicoboxil: Patients treated with ointments containing 2.5% nicoboxil alone
- Nonivamide: Patients treated with ointments containing 0.4% nonivamide alone
- Nicoboxil/Nonivamide: Patients treated with ointments containing a combination of 2.5% nicoboxil and 0.4% nonivamide
Period: Overall Study
Arm/Group | Placebo | Nicoboxil | Nonivamide | Nicoboxil/Nonivamide
Started | 204 | 201 | 198 | 202
Completed | 118 | 139 | 152 | 169
Not Completed | 86 | 62 | 46 | 33
Not completed — Adverse Event | 1 | 0 | 9 | 13
Not completed — Lack of Efficacy | 84 | 60 | 35 | 15
Not completed — Protocol Violation | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 2
Not completed — Other reasons than stated above | 1 | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Population: Patients from Treated Set (TS): Patients who were randomised and who used at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Nicoboxil | Nonivamide | Nicoboxil/Nonivamide | Total
Number analyzed (Participants) | 204 | 201 | 198 | 202 | 805
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (13.27) | 40.4 (13.06) | 42.2 (13.53) | 40.2 (14.31) | 40.5 (13.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 94 | 91 | 103 | 100 | 388
  Male | 110 | 110 | 95 | 102 | 417

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity Difference (PID) Between Pre-dose Baseline and 8hours After First Application
Description: Pain intensity (PI) was assessed on a 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst pain possible) at pre-dose baseline and 0.5, 1, 2, 3, 4, 6 and 8 hours after first ointment application. Means were adjusted for centre effect and baseline value.
Time Frame: Baseline and 8 hours after first ointment application
Population: Patients from the Full Analysis Set (FAS): all randomised patients who used at least 1 dose of study medication and provided any post-treatment data for the pain intensity difference within 8 hours after first application.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nicoboxil | Nonivamide | Nicoboxil/Nonivamide
Number analyzed (Participants) | 204 | 201 | 198 | 202
units on a scale | -1.049 (0.106) | -1.428 (0.109) | -2.252 (0.141) | -2.410 (0.138)
Statistical Analysis 1: Comparison: Placebo vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p < 0.0001, Restricted Maximum Likelihood (REML) — Model included the fixed, categorical effects of treatment, centre, time, treatment-by-time interaction and the continuous covariate of baseline PI; REML based on Repeated Measures Model, using all Available Longitudinal Pain Intensity Observations at each Post-baseline time up to 8 hours; Mean Difference (Final Values) = -1.362, 95% CI 2-sided [-1.699 to -1.025], Standard Error of Mean 0.171
Statistical Analysis 2: Comparison: Nicoboxil vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p < 0.0001, Restricted Maximum Likelihood (REML) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.983, 95% CI 2-sided [-1.324 to -0.642], Standard Error of Mean 0.173
Statistical Analysis 3: Comparison: Nonivamide vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p = 0.4171, Restricted Maximum Likelihood (REML) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.158, 95% CI [-0.541 to 0.225], Standard Error of Mean 0.195

2. Secondary Outcome: Pain Intensity Difference (PID) Between Pre-dose Baseline and 4 Hours After First Application
Description: Pain intensity was assessed on a 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst pain possible) at pre-dose baseline and 0.5, 1, 2, 3 and 4 hours after first ointment application. Means were adjusted for centre effect and baseline value.
Time Frame: Baseline and 4 hours after first ointment application
Population: Patients from FAS.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nicoboxil | Nonivamide | Nicoboxil/Nonivamide
Number analyzed (Participants) | 204 | 201 | 198 | 202
units on a scale | -0.650 (0.077) | -0.968 (0.091) | -1.641 (0.110) | -1.699 (0.109)
Statistical Analysis 1: Comparison: Placebo vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p < 0.0001, Restricted Maximum Likelihood (REML) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.049, 95% CI [-1.305 to -0.793], Standard Error of Mean 0.130
Statistical Analysis 2: Comparison: Nicoboxil vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p < 0.0001, Restricted Maximum Likelihood (REML) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.731, 95% CI [-1.003 to -0.459], Standard Error of Mean 0.138
Statistical Analysis 3: Comparison: Nonivamide vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p = 0.7037, Restricted Maximum Likelihood (REML) — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.058, 95% CI [-0.356 to 0.241], Standard Error of Mean 0.152

3. Secondary Outcome: Difference Between Baseline Pain Intensity and Average Pain Intensity on the Last Individual Treatment Day
Description: Average pain intensity was assessed in the evening of days 1, 2, 3 and 4 on a 11-point numerical rating scale ranging from 0 (no pain) to 10 (worst pain possible). The last individual treatment day is the last day with diary-recorded ointment application. Means were adjusted for centre effect and baseline value.
Time Frame: Baseline and 1 to 4 days
Population: Patients from FAS with evaluable data for the pain intensity at baseline and for the avarage pain intensity on the last individual treatment day.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Nicoboxil | Nonivamide | Nicoboxil/Nonivamide
Number analyzed (Participants) | 200 | 200 | 198 | 199
units on a scale | -1.884 (0.160) | -2.371 (0.160) | -3.074 (0.161) | -3.540 (0.159)
Statistical Analysis 1: Comparison: Placebo vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p < 0.0001, ANCOVA; The statistical model included baseline PI, centre, and treatment; Mean Difference (Final Values) = -1.655, 95% CI [-2.064 to -1.247], Standard Error of Mean 0.208
Statistical Analysis 2: Comparison: Nicoboxil vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p < 0.0001, ANCOVA; The statistical model included baseline PI, centre, and treatment; Mean Difference (Final Values) = -1.169, 95% CI [-1.578 to -0.759], Standard Error of Mean 0.209
Statistical Analysis 3: Comparison: Nonivamide vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p = 0.0259, ANCOVA; The statistical model included baseline PI, centre, and treatment; Mean Difference (Final Values) = -0.466, 95% CI [-0.875 to -0.056], Standard Error of Mean 0.209

4. Secondary Outcome: Patient Assessment of Efficacy on the Last Individual Treatment Day
Description: Patient assessment of efficacy was assessed on a 4-point verbal rating scale (VRS, 0 = 'poor', 1 = 'fair', 2 = 'good', 3 = 'very good' relief of the patients' low back pain) in the evening of days 1, 2, 3 and 4. The last individual treatment day is the last day with diary-recorded ointment application
Time Frame: 1 to 4 days
Population: Patients from FAS.
Measure: Number; unit: participants
Arm/Group | Placebo | Nicoboxil | Nonivamide | Nicoboxil/Nonivamide
Number analyzed (Participants) | 204 | 201 | 198 | 202
participants
  Very good | 9 (0.160) | 19 (0.160) | 34 (0.161) | 50 (0.159)
  Good | 47 | 67 | 85 | 88
  Fair | 22 | 20 | 27 | 20
  Poor | 125 | 94 | 52 | 42
  Missing | 1 | 1 | 0 | 2
Statistical Analysis 1: Comparison: Placebo vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The logistic regression model included baseline PI, centre, and treatment; Odds Ratio (OR) = 7.385, 95% CI [4.943 to 11.032] — Odds Ratio was calculated by Nicoboxil/Nonivamide : Placebo. Odds ratios > 1 favour Nicoboxil/Nonivamide
Statistical Analysis 2: Comparison: Nicoboxil vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p < 0.0001, Regression, Logistic; The logistic regression model included baseline PI, centre, and treatment; Odds Ratio (OR) = 3.620, 95% CI [2.469 to 5.308] — Odds Ratio was calculated by Nicoboxil/Nonivamide : Nicoboxil. Odds ratios > 1 favour Nicoboxil/Nonivamide
Statistical Analysis 3: Comparison: Nonivamide vs Nicoboxil/Nonivamide; Test type: Superiority or Other; p = 0.0129, Regression, Logistic; The logistic regression model included baseline PI, centre, and treatment; Odds Ratio (OR) = 1.594, 95% CI [1.104 to 2.303] — Odds Ratio was calculated by Nicoboxil/Nonivamide : Nonivamide. Odds ratios > 1 favour Nicoboxil/Nonivamide

ADVERSE EVENTS:
Time Frame: Up to 4 days
Groups:
- Nicoboxil/Nonivamide: Patients treated with ointments containing a combination of 2.5% nicoboxil and 0.4% nonivamide alone
Arm/Group | Placebo | Nicoboxil | Nonivamide | Nicoboxil/Nonivamide
Serious Adverse Events (participants affected / at risk) | 0/204 | 0/201 | 1/198 | 0/202
Other Adverse Events (participants affected / at risk) | 0/204 | 0/201 | 0/198 | 0/202
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=204) | Nicoboxil (N=201) | Nonivamide (N=198) | Nicoboxil/Nonivamide (N=202)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.